CLINICAL TRIAL: NCT03442465
Title: Assessment of Healing and Function After Surgical Reconstruction for Neoplasms Involving Bone
Brief Title: Assessment of Healing and Function After Reconstruction Surgery for Bone Sarcomas
Status: Recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 18-014
Record Dates: First submitted 2018-02-15; First posted 2018-02-22 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Bone Sarcoma; Osteosarcoma; Chondrosarcoma; Ewing's Sarcoma; Osseous Sarcoma; Bone Neoplasm
Keywords: 18-014; Memorial Sloan Kettering Cancer Center
MeSH Terms: conditions — Bone Neoplasms; Osteosarcoma; Chondrosarcoma; Sarcoma, Ewing | interventions — Weight-Bearing; Range of Motion, Articular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Regenerative Osseous Surgery: Participants undergoing osseous reconstructive surgery (RegOS) for bone neoplasm. Study visits for post-op assessments will be annually after month-36.
  Interventions: Behavioral: Toronto Extremity Salvage Score; Behavioral: Musculoskeletal Tumor Society Score; Behavioral: Timed Get Up and Go Test; Diagnostic Test: Orthogonal Radiographs; Diagnostic Test: Weight Bearing for lower extremities only; Diagnostic Test: Range of Motion
- Other Reconstructive Surgery: Participants undergoing other reconstructive surgery for bone neoplasm. Study visits for post-op assessments will be annually after month-36.
  Interventions: Behavioral: Toronto Extremity Salvage Score; Behavioral: Musculoskeletal Tumor Society Score; Behavioral: Timed Get Up and Go Test; Diagnostic Test: Orthogonal Radiographs; Diagnostic Test: Weight Bearing for lower extremities only; Diagnostic Test: Range of Motion

INTERVENTIONS:
Behavioral: Toronto Extremity Salvage Score — Participant-reported outcome score. For lower extremities, this is a 33 item questionnaire containing 32 5 point Likert scale items and 1 open ended response item. For upper extremities, this is a 31 item questionnaire containing 31 5 point Likert scale items and 1 open ended response item. Individual item responses range from 1-5 with higher values indicating a task is easier to complete. A total questionnaire score can also be calculated by taking the sum of the scores minus the number of total items answered, and dividing this by the maximum possible score based on the number of items answered. This results in a range from 0 -100% with higher values indicating greater ability to complete tasks 31. This scoring allows for the fact that some items may not be answered if they do not apply to an individual. It is anticipated that it will take 20 minutes to complete. Scores for the lower extremity and upper extremity may be combined, but we intend to treat them separately for analysis.
  Other Names: TESS
Behavioral: Musculoskeletal Tumor Society Score — Clinician-reported global score. For lower extremities, this is a 6 item questionnaire containing 6 point Likert scale items which cover pain, function, emotional acceptance, walking ability, gait, and necessary support. Individual item scores range from 0-5 with higher values indicating greater function, less pain, or more positive emotional acceptance. For upper extremities, this is a 6 item questionnaire containing 6 point Likert scale items which cover pain, function, emotional acceptance, hand positioning, manual dexterity, and lifting ability. Individual item scores range from 0-5 with higher values indicating greater function, less pain, or more positive emotional acceptance. A total questionnaire score which is defined as the sum of the individual items divided by the maximum possible score (5 times the number of items) may also be computed. It is represented as a percentage from 0 - 100%.
  Other Names: MSTS 3
Behavioral: Timed Get Up and Go Test — Validated functional measurement, for lower extremities only. The patient is observed and timed while s/he rises from an arm chair, walks 3 meters, turns, walks back, and sits down again. The test predicts the patient's ability to go outside alone safely and quantifies functional mobility. The test requires no special equipment and will take less than one minute to complete.
Diagnostic Test: Orthogonal Radiographs — The distance of bone transport is measured, accounting for calibration of the radiographs. The presence of bone regenerate between the transported segment is determined by the presence of continuous calcified callus from the proximal segment to the distal segment. Each of the orthogonal radiographs is used to visualize two cortices: the AP radiographs visualizes the medial and lateral cortices and the lateral radiograph measures the anterior and posterior cortices. Each continuous calcified cortex is counted with a range from 0 to 4 cortices intact.
  Other Names: Radiographic Assessments
Diagnostic Test: Weight Bearing for lower extremities only — As part of the current standard of care, patients are asked to stand on a scale with the affected lower extremity on the scale and the unaffected extremity on a block which is level with the scale. The patient is asked to place as much weight as possible on the affected extremity and this weight Is recorded. Each patient's total weight is then measured and the percent of weight bearing is calculated as the amount of weight bearing over the total body weight.
Diagnostic Test: Range of Motion — As part of the current standard of care, the joints of the affected extremity are assessed for passive range of motion at each follow up visit by the clinician. If surgery is on the femur, the hip and knee joints are assessed for range of motion. Whereas for the tibia, the knee and ankle joints are assessed. These assessments would be measured using a goniometer placed alongside the extremity and recorded for each direction of movement. Hip range of motion includes flexion, extension, abduction, internal rotation and external rotation. Knee range of motion includes flexion and extension. Ankle range of motion includes dorsiflexion and plantarflexion.

SUMMARY:
The purpose of this study is to look at the amount of function that returns in participants that have reconstruction with bone graft or artificial device and in participants who have tumor surgery plus regenerative osseous surgery.

The study will look at the level of function for a period of 3 years after the surgery. Another purpose of this study is to look at how well the bone heals in participants undergoing regenerative surgery

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing reconstructive surgery for neoplasms involving bone on the orthopaedic surgery service at MSK
* Current or prior history of primary neoplasms involving osseous structures, including all subtypes
* Confirmation of diagnosis that has been performed by the MSK's Department of Pathology via direct review of tissue/slides
* Patients must read and understand English
* Age >/=4
* Patients must read and understand English

Exclusion Criteria:

* Patients that weight <17 kilograms

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All participants who undergo osseous reconstructive surgery at Memorial Sloan Kettering Cancer Center
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-02-14 (Actual); Primary Completion 2026-02-14 (Estimated); Study Completion 2026-02-14 (Estimated)

PRIMARY OUTCOMES:
Early recovery level | 1 year from surgery
  The primary objective is to assess early recovery level of function of all participants undergoing reconstructive surgery after resection of osseous neoplasms. The early time frame is considered at one year from the neoplasm resection surgery.
Mid-recovery level | 3 years from surgery
  The primary objective is to assess mid-recovery level of function of all participants undergoing reconstructive surgery after resection of osseous neoplasms. The mid-recovery time frame is considered at one year from the neoplasm resection surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Prince, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (3):
- United States (3):
  - Memorial Sloan Kettering Monmouth (Consent and Followup), Middletown, New Jersey
  - Memorial Sloan Kettering Westchester (Consent and Followup), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://mskcc.org